CLINICAL TRIAL: NCT05200897
Title: Safety and Effects of Cefaly on Mild Cognitive Impairment With Insomnia and Exploration of Structural and Functional Connectivity Changes
Brief Title: Transdermal Trigeminal Electrical Neuromodulation on Mild Cognitive Impairment With Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Yoo Hyun Um, Clinical Assistant Professor, Saint Vincent's Hospital, Korea
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VC21DNSI0029
Record Dates: First submitted 2021-12-05; First posted 2022-01-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Insomnia; Alzheimer Disease; Mild Cognitive Impairment; Amyloid
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Amyloid positive mild cognitive impairment+ BDNF met carrier (Experimental): Transdermal trigeminal electrical modulation for 3 months
  Interventions: Device: Transdermal trigeminal electrical neuromodulation(Cefaly)
- Amyloid positive mild cognitive impairment+ BDNF Val/Val (Experimental): Transdermal trigeminal electrical modulation for 3 months
  Interventions: Device: Transdermal trigeminal electrical neuromodulation(Cefaly)
- Amyloid negative mild cognitive impairment+ BDNF met carrier (Experimental): Transdermal trigeminal electrical modulation for 3 months
  Interventions: Device: Transdermal trigeminal electrical neuromodulation(Cefaly)
- Amyloid negative mild cognitive impairment+ BDNF Val/Val (Experimental): Transdermal trigeminal electrical modulation for 3 months
  Interventions: Device: Transdermal trigeminal electrical neuromodulation(Cefaly)

INTERVENTIONS:
Device: Transdermal trigeminal electrical neuromodulation(Cefaly) — The Cefaly device delivers electrical micro-impulses through a self-adhesive electrode which is placed over the participant's forehead, where the supratrochlear and supraorbital branches of the ophthalmic division of the trigeminal nerve are located. Rectangular, biphasic impulses with an electrical mean equal to zero are transmitted. The impulse width is 250μs, frequency is 60Hz, and the maximum intensity of 16mA is over 14 minutes

SUMMARY:
This study aims to validate the safety and impact of transdermal trigeminal electrical neuromodulation(Cefaly) on mild cognitive impairment patients with insomnia on brain functional and structural connectivity as well as sleep parameters evidenced by polysomnography and sleep surveys, with consideration for amyloid positivity and brain-derived neurotrophic factor .

DETAILED DESCRIPTION:
This study aims to validate the safety and impact of transdermal trigeminal electrical neuromodulation(Cefaly) on mild cognitive impairment patients with insomnia on brain functional and structural connectivity as well as sleep parameters evidenced by polysomnography and sleep surveys, with consideration for amyloid positivity and brain-derived neurotrophic factor . A 3-month intervention with transdermal trigeminal electrical neuromodulation will be implemented and sleep surveys, polysomnography and brain MRI will be attained both at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild cognitive impairment by modified Peterson's criteria
* Identified as amyloid positive by amyloid PET result
* Insomnia severity index of more than 15 or diagnosed with insomnia disorder by Diagnostic Statistical Manual-5

Exclusion Criteria:

* Subjects with active psychiatric or neurological disorders
* Unstable medical conditions (Myocardial infarction, cerebral infarction, congestive heart failures etc.)
* Moderate to severe obstructive sleep apnea (apnea hypopnea index of more than 15), rapid eye movement disorder, narcolepsy
* On regular hypnotic medication (can enroll if there was 2-week wash out period)
* Currently receiving or having a past history of cognitive behavioral therapy for insomnia
* Patients who received transcranial magnetic stimulation (TMS), transcranial direct current stimulation, within 2 weeks before enrollment
* Who are on cognitive enhancers (choline alfoscerate, acetylcarnitine, acetylcholinesterase inhibitors, NMDA receptor antagonist)
* History of cerebral infarction or Parkinson's disease
* History of facial or brain trauma
* A subject with allergy to acrylic acid
* A subject who is sensitive to electrical devices
* A subject who are uncooperative to MRI process

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline Pittsburgh sleep quality index(PSQI) at 3 months | Post 3-month intervention
  PSQI global score of more than 5 signifies major sleep disturbance, higher scores suggesting greater sleep disturbance
Changes from Baseline Insomnia severity index(ISI) at 3 months | Post 3-month intervention
  ISI is a brief, self-rated scale that is widely used to measure insomnia severity. With seven items scored on a 0-4 scale, it only takes about 5 minutes to complete and scores of 15 or more indicates insomnia of moderate to severe severity
Changes from Baseline Epworth sleepiness scale(ESS) at 3 months | Post-3 month intervention
  ESS is a self-administered scale with eight questionnaires measuring sleepiness in daily life. Score of more than 10 signifies clinically meaningful daytime sleepiness, with higher scores indicating more severe sleepiness.
Changes from Baseline Total time in bed(TIB) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Total sleep time(TST) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Sleep efficiency(SE) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Proportion of stage 1 sleep(N1, %) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Proportion of stage 2 sleep(N2, %) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Proportion of stage 3 sleep(N3, %) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Proportion of REM sleep(R, %) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline REM sleep latency(REML) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Sleep latency(SL) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Apnea-hypopnea index(AHI) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Limb movement index(LMI) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Periodic limb movement index(PLMI) at 3 months | Post 3-month intervention
  One of polysomnography measures
Changes from Baseline Cortical thickness changes at 3 months | Post 3-month intervention
  One of neuroimaging measures
Changes from Baseline Functional connectivity measure at 3 months | Post 3-month intervention
  One of neuroimaging measures
Changes from Baseline Fractional anisotropy at 3 months | Post 3-month intervention
  One of neuroimaging measures
Changes from Baseline Mean diffusivity at 3 months | Post 3-month intervention
  One of neuroimaging measures
Changes from Baseline Verbal fluency at 3 months | Post 3-month intervention
  One of cognitive measures(subtest of CERAD-K)
Changes from Baseline Boston naming test at 3 months | Post 3-month intervention
  One of cognitive measures(subtest of CERAD-K)
Changes from Baseline Mini-mental status examination at 3 months | Post 3-month intervention
  One of cognitive measures(subtest of CERAD-K)
Changes from Baseline Word list recall at 3 months | Post 3-month intervention
  One of cognitive measures(subtest of CERAD-K)
Changes from Baseline Word list recognition at 3 months | Post 3-month intervention
  One of cognitive measures(subtest of CERAD-K)
Changes from Baseline Constructional recall at 3 months | Post 3-month intervention
  One of cognitive measures(subtest of CERAD-K)

CONTACTS AND LOCATIONS:
Overall Officials: Yoo Hyun Um, Principal Investigator — St.Vincent's Hospital, College of Medicine, Catholic University of Korea
Locations (1):
- St.Vincent's Hospital, the Catholic University of Korea, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No